CLINICAL TRIAL: NCT07335068
Title: The Effects of Exercise Snacking on Physical Fitness, Cognitive Function, and Chronic Pain in Institutionalized Older Adults: A Randomized Controlled Trial
Brief Title: Effects of Exercise Snacking on Physical Fitness, Cognition, and Pain in Institutionalized Older Adults
Acronym: EXSNAKS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ivan Patrício (Other)
Collaborators: Associação Casapiana de Solidariedade (Unknown); CIDEFES - Universidade Lusofona (Unknown)
Responsible Party: Sponsor-Investigator, Ivan Patrício, Principal Investigator, Lusofona University
Organization: Lusofona University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D1025B
Record Dates: First submitted 2026-01-04; First posted 2026-01-12 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Chronic Pain; Cognition Disorders in Old Age; Physical Fitness in Older Adults
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Snacks (Experimental): The Exercise Snacks intervention comprises two daily sessions of approximately ten minutes each, five days per week (total ≈ 100 minutes/week). Each ten-minute session consists largely of alternating one-minute bouts of activity and one-minute rest. The exercises followed a structured three-month progression. Intensity targeted at a 4 on Borg CR10 Scale "somewhat hard" with progression rules (increase repetitions, range of motion and exercise difficulty).
  Interventions: Behavioral: Exercise Snacks
- Conventional Exercise (Active Comparator): Conventional Exercise comprises two supervised 50 minutes sessions per week (total ≈ 100 minutes/week). Organized in one-minute exercise/one-minute rest intervals equal in content to the snacks but performed in longer continuous practice. The exercises followed a structured three-month progression. Intensity targeted at a 4 on Borg CR10 Scale "somewhat hard" with progression rules (increase repetitions, range of motion and exercise difficulty).
  Interventions: Behavioral: Conventional Exercise

INTERVENTIONS:
Behavioral: Exercise Snacks — Exercise snacks, defined as short bouts of gentle intermittent exercise performed twice a day
  Arms: Exercise Snacks
Behavioral: Conventional Exercise — Conventional exercise consists of longer continuous practice of structured physical activity.
  Arms: Conventional Exercise

SUMMARY:
This study aims to compare the effects of two different exercise approaches on health and well-being in older adults living in residential care facilities. One approach, called "exercise snacking," consists of short and frequent bouts of physical activity spread throughout the day, while the other involves longer, structured exercise sessions performed a few times per week.

Approximately 75 adults aged 65 years and older will be randomly assigned to one of the two exercise programs and will participate for 12 weeks. The study will examine whether exercise snacking is as effective as conventional exercise in improving physical fitness, cognitive function, chronic pain intensity, quality of life, and symptoms of anxiety and depression.

The researchers hypothesize that short, intermittent exercise sessions may provide similar or greater health benefits compared to traditional exercise programs and may represent a practical and accessible strategy to promote physical activity in older adults living in institutional settings.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 65 years
* Residence in Associação Casapiana de Solidariedade

Exclusion Criteria:

* Severe cognitive impairment (MMSE 0-10)
* Unstable medical conditions (e.g., decompensated heart failure)
* Refusal of consent
* Total inability to walk/move.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2026-01-05 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Physical Fitness Assessed by the Short Physical Performance Battery (SPPB) | Baseline and 3 months
  The Short Physical Performance Battery (SPPB) is a test of lower extremity functioning that combines scores from usual gait speed, standing balance, and chair stand tests. Scores range from 0 to 12, with higher scores indicating better physical functioning.

SECONDARY OUTCOMES:
Anxiety and depression assessed by Hospital Anxiety and Depression Scale (HADS) subscale scores | From baseline to 3 months
  HADS consists of two subscales, one measuring anxiety, with seven items, and one measuring depression, with seven items, which are scored separately. Each item was answered by the participant on a 4-point (0-3) response category so the possible scores ranged from 0 to 21 for anxiety and 0 to 21 for depression. The HADS manual indicates that a score between 0 and 7 is ''normal'', between 8 and 10 ''mild'', between 11 and 14 ''moderate'' and between 15 and 21 ''severe''.
Nordic Musculoskeletal Questionnaire (NMQ) | From baseline to 3 months
  Pain will be assessed using the Nordic Musculoskeletal Questionnaire. Participants will report as yes/no the presence of chronic pain (pain that persists or recurs more than three months) in nine body regions (neck, shoulders, elbows, wrists/hands, upper back, lower back, hips/thighs, knees, and ankles/feet). Symptom intensity in the last 7 days will be rated on a numeric scale from 0 to 10, where 0 indicates no pain and 10 indicates the worst possible pain.
The 12-Item Short-Form Health Survey (SF-12) | From baseline to 3 months
  The SF-12 includes 12 items covering eight health domains (physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional, and mental health). Responses will be scored using standard algorithms to generate two summary measures: the Physical Component Summary (PCS) and the Mental Component Summary (MCS). Scores will range from 0 to 100, with higher scores indicating better health-related quality of life. Outcomes will be reported as mean PCS and MCS scores.
Mini-Mental State Examination (MMSE) | From baseline to 3 months
  Cognitive function will be assessed using the MMSE, a standardized interviewer-administered screening tool. The MMSE will evaluate orientation, attention, memory, language, and visuospatial abilities. Total scores will range from 0 to 30, with higher scores indicating better cognitive function. Cognitive impairment will be defined according to education-adjusted cut-off scores, as follows: illiterate participants ≤15 points; participants with 1 to 11 years of education ≤22 points; and participants with more than 11 years of education ≤27 points.